CLINICAL TRIAL: NCT07313150
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of QLS7305 Following Subcutaneous Administration in Healthy Chinese Participants.
Brief Title: A Phase I Trial of Subcutaneous QLS7305 in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLS7305-101
Record Dates: First submitted 2025-11-14; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers - Male and Female
Keywords: QLS7305; Double-stranded small interfering ribonucleic acid (siRNA) targeting complement; First-in-human; C3; SAD; MAD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLS7305 (Experimental): QLS7305 Injection
  Interventions: Drug: QLS7305 Injection
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: QLS7305 Injection — QLS7305 Injection
  Other Names: QLS7305
  Arms: QLS7305
Drug: Placebo Control — The placebo is a sterile solution that matches the appearance, volume, and packaging of the QLS7305 injection. It contains no active pharmaceutical ingredient and is administered subcutaneously following the same dosing schedule as the active comparator (single or multiple doses).
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and preliminary characteristics of the investigational drug QLS7305 in healthy adult participants in China. The main questions it aims to answer are:

What is the safety and tolerability profile of single and multiple subcutaneous doses of QLS7305 in healthy adults? What are the pharmacokinetic (PK) characteristics of QLS7305 and its major metabolites? What are the pharmacodynamic (PD) effects of QLS7305 on the complement system (e.g., serum C3 levels and complement activity)? Does QLS7305 induce an immunogenic response (anti-drug antibodies)? What is the effect of QLS7305 on the QTc interval? Investigators will compare different dose levels of QLS7305 to a placebo group to see the effects on safety, tolerability, and the measured parameters.

Participants will:

Be enrolled in one of two parts of the study:

Part A (Single Ascending Dose): Receive a single dose of QLS7305 or placebo. Part B (Multiple Ascending Dose): Receive multiple doses of QLS7305 or placebo (doses selected based on Part A results).

Receive prophylactic antibiotics (Penicillin V) after the first dose until their serum complement C3 level recovers, as a safety precaution.

Undergo close safety monitoring throughout the study, including a follow-up period of up to 337 days to ensure safety parameters return to acceptable levels.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of QLS7305 Injection subcutaneously administered to healthy adults. The secondary objectives are to evaluate the pharmacokinetic (PK) characteristics, the pharmacodynamic (PD) characteristics, the immunogenicity and the effect of subcutaneous injection of QLS7305 injection on QTc interval in healthy adult participants.

This study consists of two parts:

* Part A (SAD): This part employs a randomized, double-blind, placebo-controlled design. It is planned to include 5 sequential dose groups (50 mg, 100 mg, 200 mg, 400 mg, and 800 mg). A total of 36 participants are planned: 4 participants in the first dose group and 8 participants in each subsequent dose group. Within each dose group, participants will be randomized in a 3:1 ratio to receive a single dose of either QLS7305 or placebo. Dose escalation between dose groups will proceed sequentially based on the review of safety, tolerability, and PK/PD data by the SMC. The SMC may adjust the dose levels and decide on the enrollment strategy for the highest cohort (e.g., staggered enrollment) based on participant safety. The study may be terminated early if a dose is deemed intolerable or if the study objectives are met.
* Part B (MAD): This part will also use a randomized, double-blind, placebo-controlled design. It is planned to include 2 to 3 dose groups, with 8 participants in each dose group randomized 3:1 to receive QLS7305 or placebo. The specific dose levels and dosing regimen (e.g., on Day 1 and Day 29) for Part B will be determined by the SMC based on the cumulative data from Part A.

Participants will be screened from Day -77 to Day -2. After providing informed consent, participants will receive vaccinations against Neisseria meningitidis and Streptococcus pneumoniae at least two weeks prior to dosing. Eligible participants will be admitted to the clinic on Day -1 for baseline assessments. Dosing will occur on Day 1 (for both parts) and additionally on Day 29 (for Part B). Intensive safety and PK assessments will be performed. Participants will receive prophylactic antibiotic treatment (e.g., Penicillin V) post-dose, which may be discontinued based on the investigator's assessment of serum complement C3 levels and safety risk.

A long-term follow-up period of up to Day 337 post-dose is planned to monitor safety, PD markers (C3, CP, AP), and immunogenicity. Participants with suppressed complement levels at Day 169 will undergo additional follow-up every 8 weeks until recovery (or until Day 337). After Day 337, the unblinded physician may arrange for further monitoring of specific participants if complement levels remain below predefined recovery thresholds.

ELIGIBILITY:
Inclusion Criteria:

Aged between 18 and 55 years (inclusive) Physical examination, vital signs, laboratory tests, 12-lead ECG, and imaging findings are within normal ranges.

Body weight ≥50 kg for males and ≥45 kg for females, with a BM) between 18.0 and 28 kg/m² (inclusive).

Willing or has complied with the administration of meningococcal and pneumococcal vaccines as required by the protocol.

No plan to donate sperm or ova, no pregnancy plan, and voluntarily agrees to use effective contraception methods from the signing of the ICF until 12 months after administration of the investigational product.

Able to understand and comply with the study procedures, voluntarily participate in the trial, and provide written informed consent.

Exclusion Criteria:

History of food or drug allergy, and/or known allergy to GalNAc. History of definite infection with encapsulated bacteria within 6 months prior to screening.

History of recurrent or chronic infection within 3 months prior to screening. Presence or suspicion of active viral, bacterial, fungal, or parasitic infection within 1 month prior to baseline.

Any disease at screening that, in the investigator's judgment, could affect the study data.

History of malignancy. Any condition that may affect drug absorption. History of splenectomy or congenital asplenia. History of congenital or acquired complement deficiency or disorder. History of allergic diseases (e.g., allergic asthma, allergic rhinitis).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of TEAEs | 337 days

SECONDARY OUTCOMES:
Plasma and urine concentrations of QLS7305 | 337 days
Relationship between plasma concentration of QLS7305 and the change in QTc interval. | D3

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Jing, Professor, Principal Investigator — Huashan Hospital

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data that underlie the results reported in the primary publication (for the primary and secondary endpoints).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 12 months after the primary publication and ending 5 years after the end of the study.
Access Criteria: Individual participant data that underlie the results reported in this publication, after de-identification (text, tables, figures, and appendices) will be available. Proposals should be directed to jing16.wang@qilu-pharma.com. To gain access, data requestors will need to sign a data access agreement.